CLINICAL TRIAL: NCT05471128
Title: MRI Fusion Biopsy vs. Micro-Ultrasound Guided Biopsy for the Detection of Clinically Significant Prostate Cancer
Brief Title: MRI Fusion Biopsy vs. Micro-Ultrasound Guided Biopsy
Acronym: OU-SCC-PROBX
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: OU-SCC-PROBX; IRG-19-142-01 (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2022-07-13; First posted 2022-07-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Standard of Care Biopsy — Patients will be evaluated with multiparametric MRI prostate followed by ExactVu micro-ultrasound to identify target lesions all of which will be biopsied by the examiner

SUMMARY:
The purpose of this study is to find out how best to detect clinically significant lesions of prostate cancer by using micro-ultrasound technology (ExactVu) and by multiparametric magnetic-resonance imaging (mpMRI).

DETAILED DESCRIPTION:
This is a pilot clinical trial with 30 patients with either: 1) suspected prostate cancer (based on elevated PSA or abnormal digital rectal exam (DRE), or 2) known low-risk prostate cancer being managed with active surveillance.

Enrolled patients will undergo MRI fusion biopsy and standard-template 12 core TRUS biopsy as the standard-of-care. Patients will also undergo micro-ultrasound evaluation and targeted biopsy if lesions are identified. Detection rates of clinically significant lesions by ExactVu and by MRI will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to undergo biopsy and with one of the following:

   * Men with suspicion of prostate cancer
   * Men on active surveillance
2. Age ≥18 [30]
3. Have available multiparametric prostate MRI
4. Able to provide written, informed consent
5. No significant medical illness which in the opinion of the Investigator would preclude entry to study procedures
6. Be willing and able to comply with scheduled visits

Exclusion Criteria:

1. Previously confirmed prostate cancer diagnosis with Grade Group >= 2
2. Unable to undergo prostate biopsy
3. Prostate MRI unable to be evaluated using the PI-RADS v2 criteria
4. Men with contraindication for MRI or a prostate biopsy
5. Prostate biopsy within 8 weeks prior to mpMRI.
6. Any history of prostate treatment

Ages: 18 Years to 99 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: The study population will cover all races, including socioeconomically disadvantaged minorities, that have been diagnosed with prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Detection Rate | 2 years
  To compare the detection rates of clinically significant prostate cancer lesions by ExactVu micro-ultrasound and by MRI-fusion
Feasibility of ExactVu | 2 years
  To determine the feasibility of using ExactVu micro-ultrasounds to screen for prostate cancer in socioeconomically disadvantaged populations with limited access to care. Feasibility is measured by the percentage of patients that successfully undergo the study procedures.

SECONDARY OUTCOMES:
Predictive Performance Measures | 2 years
  To evaluate the sensitivity of ExactVu micro-ultrasound method and MRI-fusion method in detection of prostate cancer
Predictive Performance Measures | 2 years
  To evaluate the negative predictive value of ExactVu micro-ultrasound method and MRI-fusion method in detection of prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McIntosh, MD, Principal Investigator — University of Oklahoma Stephenson Cancer Center
Locations (1):
- University of Oklahoma Health Sciences Center, Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No